CLINICAL TRIAL: NCT03001154
Title: Virtual Reality Exposure Therapy for Speech Anxiety Using Commercial Hardware and Software
Acronym: VRETORIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRetorik
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Social Phobia; Anxiety; Behavior Therapy
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-session VRET face-to-face (Experimental): One-session Virtual Reality Exposure Therapy led by therapist (face-to-face), followed by a 4-week therapist-guided Internet-administered progressive maintenance program.
  Interventions: Behavioral: Face-to-face Virtual Reality Exposure Therapy
- Waiting-list, then Internet-administered VRET (Experimental): 4-week waiting list, followed by therapist-guided, Internet-administered VRET with a 4-week progressive maintenance program.
  Interventions: Behavioral: Internet-administered Virtual Reality Exposure Therapy; Other: Waiting-list

INTERVENTIONS:
Behavioral: Face-to-face Virtual Reality Exposure Therapy — In session, systematic, hierarchical exposure to feared stimuli with therapist.
  Arms: One-session VRET face-to-face
Behavioral: Internet-administered Virtual Reality Exposure Therapy — Therapist-guided, Internet-administered Virtual Reality Exposure Therapy self-help program
  Arms: Waiting-list, then Internet-administered VRET
Other: Waiting-list — Weekly assessments of public speaking
  Arms: Waiting-list, then Internet-administered VRET

SUMMARY:
Virtual Reality Exposure Therapy (VRET) is an efficacious treatment of fear and anxiety, but because of the high financial costs and technical complexity of the past generation of VR hardware, there has been no large-scale implementation of this promising treatment. The present study will investigate whether off-the-shelf, commercial VR hardware and software can be used as stimuli material to conduct in-session exposure therapy for speech anxiety. The study will recruit n=25+25 participants from the general public suffering from substantial speech anxiety, who will be randomized to either a waiting-list, or one-session VRET with a therapist, followed by four weeks of a progressive maintenance program encouraging in-vivo exposure. The waiting-list group will then receive an Internet-delivered VRET treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Substantial public speaking anxiety
* Have access to VR-compatible smartphone (including Internet)
* Can travel to Stockholm University for treatment on one occasion
* Can speak and understand sufficient Swedish

Exclusion Criteria:

* Deficits in sight or balance impacting the VR-experience
* A severe psychiatric disorder better treated elsewhere, including current major depression, alcohol or drug abuse, bipolarity, psychosis or similar
* Active psychopharmacological treatment, unless stable for last 3 months
* Other ongoing psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Public Speaking Anxiety Scale | Change from baseline: Week 0, 1, 2, 3, 4, 5 and 21
  Self-rating of public speaking anxiety

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale Self-Report | Change from baseline: Week 0, 5 and 21
  Self-rating of general social anxiety
Brief Fear of Negative Evaluation Scale | Change from baseline: Week 0, 5 and 21
  Self-rating of fear of negative evaluation
Patient Health Questionnaire 9-item | Change from baseline: Week 0, 5 and 21
  Self-rating of depressive symptoms
Generalized Anxiety Disorder 7-item | Change from baseline: Week 0, 5 and 21
  Self-rating of general anxiety symptoms
Brunnsviken Brief Quality of life scale | Change from baseline: Week 0, 5 and 21
  Self-rating of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided